CLINICAL TRIAL: NCT06066541
Title: Social Norms, Messengers, and Processing Fluency to Increase Hypertension Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Humana Inc. (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023p002222; P30AG064199 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Medication Adherence; Hypertension
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Scorecard (Active Comparator): Participants randomized to this arm will receive a scorecard from Humana reporting patients' medication adherence using a "refill score." Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Interventions: Behavioral: Scorecard
- Scorecard + Social norms (Experimental): Participants randomized to this arm will receive the Arm 1 scorecard plus dynamic social norms messaging (noting the proportion of Humana members improving their medication refill scores). Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Interventions: Behavioral: Scorecard; Behavioral: Social norms
- Scorecard + Messenger effects (Experimental): Participants randomized to this arm will receive the Arm 1 scorecard, coming from the trusted messenger of a Humana-identified pharmacist taking the same medication. Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Interventions: Behavioral: Scorecard; Behavioral: Messenger effects
- Processing fluency (Experimental): Participants randomized to this arm will receive a modified scorecard increasing processing fluency through a visual metaphor of "closing the ring." Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Interventions: Behavioral: Processing fluency
- Processing fluency + Social norms (Experimental): Participants randomized to this arm will receive the Arm 4 processing fluency scorecard plus dynamic social norms messaging. Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Interventions: Behavioral: Social norms; Behavioral: Processing fluency
- Processing fluency + Messenger effects (Experimental): Participants randomized to this arm will receive the Arm 4 processing fluency scorecard coming from the trusted messenger of a Humana-identified pharmacist taking the same medication. Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Interventions: Behavioral: Messenger effects; Behavioral: Processing fluency
- Usual care (No Intervention): Participants randomized to this arm will not receive any mailed message.

INTERVENTIONS:
Behavioral: Scorecard — Participants will be mailed a scorecard from Humana reporting patients' medication adherence using a "refill score."
  Arms: Scorecard; Scorecard + Messenger effects; Scorecard + Social norms
Behavioral: Social norms — Participants will be mailed a dynamic social norms messaging (noting the proportion of Humana members improving their medication refill scores).
  Arms: Processing fluency + Social norms; Scorecard + Social norms
Behavioral: Messenger effects — Participants will be mailed a scorecard coming from the trusted messenger of a Humana-identified pharmacist taking the same medication.
  Arms: Processing fluency + Messenger effects; Scorecard + Messenger effects
Behavioral: Processing fluency — Participants will be mailed a modified scorecard increasing processing fluency through a visual metaphor of "closing the ring."
  Arms: Processing fluency; Processing fluency + Messenger effects; Processing fluency + Social norms

SUMMARY:
Medicare Advantage beneficiaries ages 65-79 and insured by Humana with at least two unique fills of hypertension medication within the 2023 calendar year and adherence level between 60 and 85% will be identified using Humana Medicare Advantage claims data. Individuals meeting these inclusion criteria will be included and, with an institutional review board approved waiver of informed consent, will be randomized to one of 6 mailed messages or control (no message). The messages will be sent by Humana and use different behavioral techniques (social norms, messenger effects, and/or processing fluency) providing their medication refill score. Humana will send a second message within 60 days of the first message noting any changes in the refill score.

The primary outcome will be the average end-of-year adherence in each arm. A secondary outcome will be the proportion of study participants with end-of-year adherence greater than or equal to 80%. The study team's hypothesis is that messages using dynamic social norms, messenger effects, and processing fluency in combination will more effectively increase average end-of-year adherence level compared to usual care.

Humana will conduct all study participant outreach and data analyses, which will be performed using routinely collected insurance claims data. Regulatory oversight is conducted using Humana's centralized institutional review board (IRB) of record. The work completed by Humana study staff is funded by Humana, Inc.

Dr. Choudhry and his colleagues (including subaward recipients ideas42 and Tuck School of Business at Dartmouth) will provide technical and subject matter expertise related to study research design and implementation, protocol design, statistical analysis, publication (abstract, poster, manuscript) preparation and/or review, and assistance throughout the peer review process including revisions and additional analyses if necessary for this project. The work completed by study staff at Brigham and Women's Hospital, ideas42, and Tuck School of Business at Dartmouth is funded by NIA.

ELIGIBILITY:
Inclusion Criteria:

* Medicare Advantage beneficiary insured by Humana
* Between the ages of 65 and 79
* Having at least two unique fills of any class of hypertension medication within the calendar year (2023).
* Adherence level (as measured by the proportion of days covered [PDC] metric) between 60% and 85%

Exclusion Criteria:

* Beneficiaries in plans which, per contractual agreements, privacy policies and rules, or legal requirements, do not participate in research

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65177 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Robertson, MPA, Principal Investigator — Ideas42; Punam Keller, PhD, MBA, Principal Investigator — Tuck School of Business at Dartmouth
Locations (1):
- Humana, Inc., Louisville, Kentucky, United States

REFERENCES:
- [Derived] Keller P, Robertson T, Kao LS, Li Y, Merrell B, Chung L, Boudreau E, James A, Esterly L, Hanken K, Choudhry NK. Incorporating Behavioral Science in Medication Adherence Communication: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2510162. doi: 10.1001/jamanetworkopen.2025.10162. PMID 40366654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomized 65,177 study participants before our study launched with recruitment starting in August 2023. We recruited in two waves (on August 18, 2023 and August 24, 2023) to ensure a sufficient sample size after adjusting for dropouts due to loss of eligibility or changes in membership.
Groups:
- Baseline Mailing (Scorecard): Participants randomized to this arm will receive a scorecard from Humana reporting patients' medication adherence using a "refill score." Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Scorecard: Participants will be mailed a scorecard from Humana reporting patients' medication adherence using a "refill score."
- Baseline Mailing + Dynamic Social Norms: Participants randomized to this arm will receive the Arm 1 scorecard plus dynamic social norms messaging (noting the proportion of Humana members improving their medication refill scores). Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Scorecard: Participants will be mailed a scorecard from Humana reporting patients' medication adherence using a "refill score."
  Social norms: Participants will be mailed a dynamic social norms messaging (noting the proportion of Humana members improving their medication refill scores).
- Baseline Mailing + Messenger Effects: Participants randomized to this arm will receive the Arm 1 scorecard, coming from the trusted messenger of a Humana-identified pharmacist taking the same medication. Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Scorecard: Participants will be mailed a scorecard from Humana reporting patients' medication adherence using a "refill score."
  Messenger effects: Participants will be mailed a scorecard coming from the trusted messenger of a Humana-identified pharmacist taking the same medication.
- Baseline Mailing + Processing Fluency: Participants randomized to this arm will receive a modified scorecard increasing processing fluency through a visual metaphor of "closing the ring." Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Processing fluency: Participants will be mailed a modified scorecard increasing processing fluency through a visual metaphor of "closing the ring."
- Processing Fluency + Dynamic Social Norms: Participants randomized to this arm will receive the Arm 4 processing fluency scorecard plus dynamic social norms messaging. Two messages will be sent during the intervention: The first message will contain the baseline refill score. The second message will note any changes in the refill score.
  Social norms: Participants will be mailed a dynamic social norms messaging (noting the proportion of Humana members improving their medication refill scores).
  Processing fluency: Participants will be mailed a modified scorecard increasing processing fluency through a visual metaphor of "closing the ring."
- No Mailing (Usual Care): Participants randomized to this arm will not receive any mailed message.
Period: Enrollment Wave 1 (August 18, 2023)
Arm/Group | Baseline Mailing (Scorecard) | Baseline Mailing + Dynamic Social Norms | Baseline Mailing + Messenger Effects | Baseline Mailing + Processing Fluency | Processing Fluency + Dynamic Social Norms | Processing Fluency + Messenger Effects | No Mailing (Usual Care)
Started (Potentially eligible Humana members randomized in first wave) | 8571 | 8571 | 8571 | 8571 | 8571 | 8571 | 8571
Completed | 8464 | 8449 | 8443 | 8461 | 8446 | 8448 | 8448
Not Completed | 107 | 122 | 128 | 110 | 125 | 123 | 123
Not completed — Excluded due to membership changes | 107 | 122 | 128 | 110 | 125 | 123 | 123
Period: Enrollment Wave 2 (August 24, 2023)
Arm/Group | Baseline Mailing (Scorecard) | Baseline Mailing + Dynamic Social Norms | Baseline Mailing + Messenger Effects | Baseline Mailing + Processing Fluency | Processing Fluency + Dynamic Social Norms | Processing Fluency + Messenger Effects | No Mailing (Usual Care)
Started (Potentially eligible Humana members randomized in second wave) | 740 | 740 | 740 | 740 | 740 | 740 | 740
Completed | 734 | 731 | 737 | 732 | 733 | 729 | 735
Not Completed | 6 | 9 | 3 | 8 | 7 | 11 | 5
Not completed — Excluded due to membership changes | 6 | 9 | 3 | 8 | 7 | 11 | 5

BASELINE CHARACTERISTICS:
Population: We randomized 65,177 study participants before our study launched with recruitment starting in August 2023. We recruited in two waves (on August 18, 2023 and August 24, 2023) to ensure a sufficient sample size after adjusting for dropouts due to loss of eligibility or changes in membership. Our final sample consisted of 64,290 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Mailing (Scorecard) | Baseline Mailing + Dynamic Social Norms | Baseline Mailing + Messenger Effects | Baseline Mailing + Processing Fluency | Processing Fluency + Dynamic Social Norms | Processing Fluency + Messenger Effects | No Mailing (Usual Care) | Total
Number analyzed (Participants) | 9198 | 9180 | 9180 | 9193 | 9179 | 9177 | 9183 | 64290
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.36 (4.11) | 71.44 (4.09) | 71.44 (4.09) | 71.33 (4.07) | 71.49 (4.10) | 71.44 (4.07) | 71.50 (4.07) | 71.4 (4.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4881 | 5005 | 5041 | 4938 | 5040 | 4967 | 4939 | 34811
  Male | 4317 | 4175 | 4139 | 4255 | 4139 | 4210 | 4244 | 29479
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5882 | 5914 | 5822 | 5837 | 5903 | 5900 | 5879 | 41137
  Black | 2229 | 2140 | 2225 | 2218 | 2114 | 2143 | 2168 | 15237
  Other | 778 | 820 | 808 | 814 | 842 | 845 | 829 | 5736
  Unknown | 309 | 306 | 325 | 324 | 320 | 289 | 307 | 2180
Refill cycle [Count of Participants; unit: Participants]
  30-day refill cycle | 1965 | 1962 | 1961 | 1977 | 1974 | 1972 | 1975 | 13786
  90-day refill cycle | 7233 | 7218 | 7219 | 7216 | 7205 | 7205 | 7208 | 50504
Low-Income Subsidy (LIS)/Dual Eligibility Status [Count of Participants; unit: Participants]
  Low-Income Subsidy (LIS) Only | 497 | 518 | 536 | 514 | 524 | 567 | 566 | 3722
  Medicaid Eligible only | 9 | 7 | 10 | 12 | 16 | 8 | 10 | 72
  LIS and Dual Eligible | 2407 | 2364 | 2289 | 2396 | 2330 | 2294 | 2296 | 16376
  No LIS/Dual Eligibility | 6285 | 6291 | 6345 | 6271 | 6309 | 6308 | 6311 | 44120
Hypertension proportion of days covered (PDC) as of selection [Mean (Standard Deviation); unit: proportion of days covered (PDC)] — proportion of days covered (PDC) in prescription insurance claims following the Medicare Star Ratings approach
  proportion of days covered (PDC) | 0.77 (0.06) | 0.77 (0.06) | 0.77 (0.06) | 0.77 (0.06) | 0.77 (0.06) | 0.77 (0.06) | 0.77 (0.06) | 0.77 (0.06)
Hypertension PDC ≥ 80% as of selection [Count of Participants; unit: Participants] | 3690 | 3615 | 3705 | 3720 | 3690 | 3650 | 3722 | 25792

OUTCOME MEASURES:

1. Primary Outcome: Average End-of-year Adherence Level
Description: The primary outcome will be the average end-of-year adherence level in each arm (as measured by the Proportion of Days Covered metric [PDC]) stratified by refill cycle and adjusting for age, sex, and race.
Time Frame: approximately 4 months
Measure: Mean (Standard Deviation); unit: proportion of days covered
Arm/Group | Baseline Mailing (Scorecard) | Baseline Mailing + Dynamic Social Norms | Baseline Mailing + Messenger Effects | Baseline Mailing + Processing Fluency | Processing Fluency + Dynamic Social Norms | Processing Fluency + Messenger Effects | No Mailing (Usual Care)
Number analyzed (Participants) | 9198 | 9180 | 9180 | 9193 | 9179 | 9177 | 9183
proportion of days covered | 0.81 (0.12) | 0.81 (0.12) | 0.81 (0.12) | 0.81 (0.12) | 0.81 (0.12) | 0.81 (0.12) | 0.81 (0.12)

2. Secondary Outcome: Proportion of Participants With End-of-year PDC≥80%
Description: As measured by the Proportion of Days Covered metric [PDC]
Time Frame: approximately 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Mailing (Scorecard) | Baseline Mailing + Dynamic Social Norms | Baseline Mailing + Messenger Effects | Baseline Mailing + Processing Fluency | Processing Fluency + Dynamic Social Norms | Processing Fluency + Messenger Effects | No Mailing (Usual Care)
Number analyzed (Participants) | 9198 | 9180 | 9180 | 9193 | 9179 | 9177 | 9183
Participants | 6518 | 6590 | 6467 | 6515 | 6558 | 6598 | 6587

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from date of participant randomization through the end of participant follow-up for all participants. Adverse event data were collected from date of participant randomization through the end of participant follow-up. Wave 1 participants were assessed for approximately 19 weeks. Wave 2 participants were assessed for approximately 18 weeks.
Description: Collection of adverse events was completed using a non-systematic assessment and was collected via self-report by Humana members.
Arm/Group | Baseline Mailing (Scorecard) | Baseline Mailing + Dynamic Social Norms | Baseline Mailing + Messenger Effects | Baseline Mailing + Processing Fluency | Processing Fluency + Dynamic Social Norms | Processing Fluency + Messenger Effects | No Mailing (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/9198 | 0/9180 | 0/9180 | 0/9193 | 0/9179 | 0/9177 | 0/9183
Serious Adverse Events (participants affected / at risk) | 0/9198 | 0/9180 | 0/9180 | 0/9193 | 0/9179 | 0/9177 | 0/9183
Other Adverse Events (participants affected / at risk) | 0/9198 | 0/9180 | 0/9180 | 0/9193 | 0/9179 | 0/9177 | 0/9183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT06066541/Prot_SAP_000.pdf